CLINICAL TRIAL: NCT03868176
Title: Phase II, Open-label, Randomized, Non-comparative Study Evaluating the Impact of Short Message Service (SMS) on Compliance With Surveillance of Patients With Germ-cell Tumors. (TEXTIS Study)
Brief Title: Study Evaluating the Impact of Short Message Service on Compliance With Surveillance of Patients With Germ-cell Tumors
Acronym: TEXTIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2018/404
Record Dates: First submitted 2019-02-04; First posted 2019-03-08 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Follow-up; Compliance, Patient; Text Messaging; Germ Cell Tumor
Keywords: surveillance; compliance; germ cell tumors; short message service
MeSH Terms: conditions — Patient Compliance; Neoplasms, Germ Cell and Embryonal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: reminder SMS before appointment: SMS before appointment detailing the date of consultation and exams to be performed before
  Interventions: Other: short message service
- Active comparator: standard of care

INTERVENTIONS:
Other: short message service — short message service
  Groups: Experimental: reminder SMS before appointment

SUMMARY:
This study will evaluate the impact of Short Message Service (SMS) on compliance with surveillance of patients with germ-cell tumors. Patients will be randomized in a 2:1 ratio to get 2 groups : (1) patients will receive reminder SMS before appointment detailing the date of consultation and exams to be performed before; (2) standard of care without SMS.

ELIGIBILITY:
Inclusion Criteria:

* Patient with germ cell tumor.
* Patient with a mobile phone.
* Patient on surveillance.

Exclusion Criteria:

* Testicular cancer without germ cell component.
* Prior history of other malignancy except for: cutaneous cancers excluding melanoma, superficial bladder tumor, localized prostate cancer with undetectable PSA.
* Cognitive condition that would preclude patient's understanding and completion of study procedures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 235 patients, with 157 in the experimental arm, with SMS sending and 78 patients in the control arm, without sending SMS.
Sampling Method: Probability Sample
Enrollment: 235 (Estimated)
Dates: Start 2019-02-28 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who report optimal compliance to surveillance | 1 year
  Optimal compliance is defined according to the following 2 parameters:
  * The patient comes to all the appointments, on the expected day, AND
  * With all the biological and imaging exams previously scheduled by the physician.

SECONDARY OUTCOMES:
Rate of patients who report intermediate compliance to surveillance | 1 year
  Intermediate compliance is defined according to the following 2 parameters:
  * The patient comes to all the appointments, but in one of the consultations, he delays his scheduled appointment of more than 3 weeks but less than 6 weeks OR
  * Missing a biological or imaging exam.
Rate of patients who report a non compliance to surveillance | 1 year
  Non compliance is defined according to the following 3 parameters:
  The patient misses a consultation, without warning, OR
  * He delays of more than 6 weeks his appointment of consultation, OR
  * At least 2 biological or imaging exams requested by the oncologist are missing from all consultations.
Patient satisfaction of sending SMS, in experimental arm | 1 year
  It is evaluated with the following question: do you find that having reminder sms for your appointments and exams is useful? evaluated on a scale of 0 to 10 (0: useless, 10: useful)
biological recurrence rate | 1 year
  Biological recurrence rate is defined by the increase in tumor markers (alpha-fetoprotein, lactic dehydrogenase, human chorionic gonadotropin).
Radiological recurrence rate | 1 year
  Radiological recurrence rate is defined according to Response evaluation criteria in solid tumors (RECIST) criteria 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Besancon, Besançon, Franche-Comté, France